CLINICAL TRIAL: NCT04621201
Title: Genomic Profiles Analysis in Children, Adolescents and Young Adult With Sarcomas (SAR-GEN_ITA): a Multicenter Prospective Study
Brief Title: Genomic Profiles Analysis in Children, Adolescents and Young Adult With Sarcomas
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Collaborators: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Professor, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: SAR-GEN_ITA
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diagnosed or Relapsed/Refractory Sarcomas
MeSH Terms: conditions — Disease; Recurrence; Sarcoma | interventions — Observation; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation and biopsy — biopsy

SUMMARY:
Bone and soft tissue sarcomas represent about 7-12% of all pediatric cancer and are a heterogeneous group of tumors arising in connective tissues embryologically derived from the mesenchyme. For some of these tumors relapse and mortality rates are still significantly high. Therefore, further studies are needed to better understand pathogenetic processes underlying sarcomas to offer new and more effective treatments. Next generation sequencing (NGS) has opened new frontiers for cancer research allowing to identify somatic or constitutional mutations known or yet unknown with the aim to better understand carcinogenesis. The establishment of the genomic profile of the tumor could also help clinicians to personalize patients treatment based on their genetic and molecular alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed Osteosarcoma, Ewing Sarcoma or Synovial Sarcoma at first diagnosis.
2. Patients with confirmed relapsed/refractory Osteosarcoma, Ewing Sarcoma or Synovial Sarcoma
3. Written informed consent signed by the patient, or parents or legal representative to perform molecular analysis of the tumor sample.
4. Patients aged ≤24 years
5. Pathological review of tumor samples.
6. Availability of fresh tumor sample from newly diagnosed or relapsed/refractory cancer and 10 ml of EDTA peripheral blood sample. Centralization of paraffin-embedded tumor sample might be optional.

Exclusion Criteria:

* 1. Known history of active HIV, HCV, or HBV infection 2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient undergoing surgery biopsy or the quality of the data.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults aged ≤ 24 years with newly diagnosed or relapsed/refractory Osteosarcoma, Ewing Sarcoma or Synovial Sarcoma.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2024-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
evaluate the genomic profiles of osteosarcoma, Ewing sarcoma and Synovial Sarcoma tumor samples in pediatric, adolescents and young adult patients at the time of diagnosis or relapse/progression | 2018-2021

CONTACTS AND LOCATIONS:
Overall Officials: Franca Fagioli, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (10):
- Italy (10):
  - AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Torino, Turin
  - Istituto Ortopedico Rizzoli, Bologna
  - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda ospedaliero-universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Istituto Nazionale Tumori, Milan
  - Presidio Ospedaliero Gaetano Pini | ASST Pini-CTO, Milan
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Istituti fisioterapici Ospitalieri - Istituto Tumori Regina Elena e Istituto Dermatologico San Gallicano, Roma
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No